CLINICAL TRIAL: NCT01639898
Title: Phase II Trial With Lenalidomide-Dexamethasone Combination in the Treatment of POEMS Syndrome.
Brief Title: POEMS Syndrome Treatment With Lenalidomide
Acronym: POEMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Ministry of Health, France (Other Government); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I10 015
Record Dates: First submitted 2012-07-05; First posted 2012-07-13 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: POEMS Syndrome
Keywords: POEMS; VEGF; Free light; lenalidomide; dexamethasone
MeSH Terms: conditions — POEMS Syndrome | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 ("2-cycles" trial) (Experimental): The "2-cycles" trial will be available to patients who can be treated by radiation or intensive treatment (75 % of cases occurring in front line); they will then undergo 2 cycles of the lenalidomide-dexamethasone combination before radiation or intensive treatment (Group 1).
  Interventions: Drug: Lenalidomide and dexamethasone
- Group 2 ( "9 cylces" Trial) (Experimental): The "9-cycles" trial will be available to all other front-line patients (25 % of front-line patients) or patients in relapse or resistant, they will undergo 9 cycles of the lenalidomide-dexamethasone combination followed by maintenance therapy with lenalidomide alone for one year (Group 2).
  Interventions: Drug: Lenalidomide and dexamethasone

INTERVENTIONS:
Drug: Lenalidomide and dexamethasone — 2 cycles of the lenalidomide-dexamethasone (Len-Dex) combination before radiation or intensive treatment
  Arms: Group 1 ("2-cycles" trial)
Drug: Lenalidomide and dexamethasone — 9 cycles of the Len-Dex combination
  Arms: Group 2 ( "9 cylces" Trial)

SUMMARY:
POEMS syndrome is a rare form of B cell dyscrasia combining a proliferation usually of plasma cells, a polyneuropathy, osteocondensing bone lesions and multiple other clinical signs. Lenalidomide appears to be particularly efficient in this pathology.

The investigators propose a phase II multicentre protocol, based on the use of lenalidomide combined with dexamethasone in patients presenting a POEMS syndrome, either de novo or resistant or in relapse.

Patients who can be treated by local radiation or intensive treatment with stem cell support will undergo 2 cycles of the lenalidomide-dexamethasone (Len-Dex) combination before radiation or intensive treatment (Group 1), the other patients will undergo 9 cycles of the Len-Dex combination (Group 2).

A biological study is coupled with this clinical protocol in order to define the best biological markers predicting clinical responses, to better understand the POEMS pathophysiological mechanisms and to set up a bank of samples which can be used to study this rare pathology.

DETAILED DESCRIPTION:
The investigators propose to simultaneously set up two Phase II therapeutic trials: Trial "2 cycles" and trial "9 cycles" (Fleming plan in one stage).

This will mean prospective multicentre studies, around a treatment with the lenalidomide-dexamethasone combination in patients suffering from POEMS syndrome either de novo, resistant or in relapse.

Both trials carried out in parallel are complementary regarding the eligibility criteria:

* Group 1: the "2-cycles" trial will be available to patients who can be treated by radiation or intensive treatment (75 % of cases occurring in front line); they will then undergo 2 cycles of the lenalidomide-dexamethasone combination before radiation or intensive treatment (Group 1).
* Group 2 : the "9-cycles" trial will be available to all other front-line patients (25 % of front-line patients) or patients in relapse or resistant, they will undergo 9 cycles of the lenalidomide-dexamethasone combination followed by maintenance therapy with lenalidomide alone for one year (Group 2).

Both these trials carried out within the same study will enable us to answer the question of potential efficacy of lenalidomide in POEMS syndrome and could enable us to draw up a new therapeutic standard.

Main objective:

Group 1: to evaluate the efficacy of the Len-Dex combination on the biological response after 2 cycles in patients with POEMS syndrome who can undergo radiation or intensive treatment.

Group 2: to evaluate the efficacy of the Len-Dex combination on the biological response in patients with POEMS syndrome who cannot be treated by radiation or intensive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from POEMS syndrome (Mayo Clinic criteria)
* Patients with a localised disease who can be treated with radiation and those with a disseminated disease and who can be treated intensively will be included in Group 1, all other patients will be included in Group 2.
* Patients aged of 18 or more
* Patients who do not show uncontrolled thrombosis
* Patients who have been duly informed and who have signed a consent form.
* Patients must respect all the lenalidomide Pregnancy Prevention Program (PPP) requirements described in appendix of the protocol.
* Patients registered with the French National Health System.

Exclusion Criteria:

* Women who are pregnant, or suspected to be pregnant or breastfeeding
* Pathology not linked with POEMS, contraindicating one of the studied drugs
* Patients suffering from a deficiency which does not allow them full understanding of the trial requirements and which could compromise proper consent from the patient and/or observance of the protocol and continuous participation in the trial.
* Prior history of malignancy other than POEMS syndrome or active other cancer or other serious illness.
* Any contraindication to Revlimid® or to one of its excipient.
* Patient with clearance creatinine < 30mL/min.
* Hepatic insufficiency
* Patient with Absolute Neutrophil count (ANC) < 1,0 x 109/L
* Patient with platelet count < 75 x 109/L
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* Instable, clinically significant ECG findings
* Known positive for HIV, or active infectious hepatitis, type A, B or C
* Patients under protection of a legal order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Biological outcome | Two months for group 1
  Decrease of monoclonal protein and serum VEGF level
Biological outcome | 2, 4 or 6 month for group 2
  Decrease of monoclonal protein and serum VEGF level

SECONDARY OUTCOMES:
Clinical response | 2 months
  Evaluation of the neurological (Overall Neuropathy Limitations Scale, Neuropsychological Impairment Scale and 10 m walking test) and other damages responses:

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud JACCARD, MD, Study Chair — CHU Limoges
Locations (11):
- France (11):
  - CHU d'Angers, Angers
  - CHU de Caen, Caen
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - Hospices Civil de Lyon, Lyon
  - Centre Léon Bérard, Lyon
  - CHU de Nantes, Nantes
  - Hôpital Saint-Louis, Paris
  - Pitié Salpétrière, Paris
  - Hôpital Necker, Paris
  - CHU de Toulouse, Toulouse